CLINICAL TRIAL: NCT01114958
Title: A Phase I / Pilot Study of Intra-Arterial Supradose Cisplatin With Simultaneous Intravenous Thiosulfate Neutralization in Patients With Primary Lung Cancer or Lung Metastases
Brief Title: Pilot Study of Intra-Arterial Cisplatin With IV Thiosulfate in Patients With Lung Cancer or Lung Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Gregory Daniels, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD 090772
Record Dates: First submitted 2010-04-28; First posted 2010-05-03 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Lung Neoplasms; Neoplasm Metastasis
Keywords: Lung cancer; Non-small cell lung cancer; Small-cell lung cancer; Lung metastases; Metastatic cancer; Stage IIIA; Stage IIIB; Stage III; Stage 3
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Cisplatin; Thiosulfates

ARMS (1):
- IA Cisplatin / IV Thiosulfate (Experimental): Single-arm study
  Interventions: Drug: Cisplatin, Thiosulfate

INTERVENTIONS:
Drug: Cisplatin, Thiosulfate — Cisplatin (150 mg/m^2) is given as an intra-arterial bolus, once, on days 2 and 9 of treatment. Thiosulfate (9 g/m^2), is given concurrently with cisplatin as an intravenous push over 15-20 minutes followed by a 6-hour intravenous infusion of thiosulfate (12 g/m^2).

SUMMARY:
This phase I study proposes the use of systemic thiosulfate rescue to allow supradose intra-arterial cisplatin delivery to lung tumors. Eligible patients would be those with at least one lung lesion large enough of characterize angiographically. All patients will first undergo a CT arteriogram of the target tumor. Patients will then receive 2 treatments on 2 consecutive weeks. The primary endpoint will be toxicity, with secondary endpoint of response as measured on week 4. This pilot study will also determine how technically feasible it is to locate the blood supply to these tumors and deliver cisplatin.

If the first 6 patients do well, 6 additional patients will be accrued for a total of 12.

ELIGIBILITY:
Inclusion Criteria:

* Primary lung cancer (any type) or dominant lung metastases from other primary cancers.
* Patients must have either measurable or evaluable disease.
* Karnofsky performance status ≥ 70%.
* Greater than 18 years of age.
* Life expectancy > 3 months.
* 3 week elapse from previous cytotoxic therapy (except for erlotinib or hormonal therapy, which can be ongoing) with side effects improved to grade 2 or less, and no prior radiotherapy to the lung.
* Adequate organ function.
* Treated brain metastases, if present, with toxicities improved to grade 2 or less.
* Willingness and ability to sign a written informed consent.

Exclusion Criteria:

* Prior radiation to the largest lesion in the lung.
* Current pregnancy or breast-feeding.
* Unwillingness or inability to practice contraception.
* Renal insufficiency.
* Comorbidities of grade 3 or greater.
* Concurrent medical or psychiatric conditions as defined by the treating physician which would preclude safe performance of study procedures or compromise the ability of the patient to consent to study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-09-03 (Actual); Primary Completion 2013-05-17 (Actual); Study Completion 2013-05-17 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events due to intra-arterial cisplatin administration | One week after treatment
  To characterize the toxicity of intra-arterial supradose cisplatin with thiosulfate rescue when delivered as two doses, one week apart, for patients with primary lung tumors and/or lung metastases.

SECONDARY OUTCOMES:
Radiographic determination of the tumor response rate in patients with primary and metastatic lung tumors treated with intra-arterial supradose cisplatin. | 4 weeks after first dose of cisplatin
Angiographic delineation of the vascular structure of primary lung tumors and lung metastases. | Once before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Daniels, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Moores Cancer Center, La Jolla, California, United States